CLINICAL TRIAL: NCT03922737
Title: Evaluation of Telehealth Follow-up Appointments Following Orthopaedic Surgery
Brief Title: Telehealth Following Orthopaedic Procedures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019Horneff
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Post-Op Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-person office visit (Active Comparator)
  Interventions: Procedure: In-person office visit
- Telehealth visit with provider (Active Comparator)
  Interventions: Procedure: Teleheath visit

INTERVENTIONS:
Procedure: In-person office visit — Post-operative visit to occur in-person with provider
  Arms: In-person office visit
Procedure: Teleheath visit — Post-operative visit to occur via telehealth software platform with provider
  Arms: Telehealth visit with provider

SUMMARY:
This study aims to evaluate the quality of care provided by a home-based teleheath program as a safe and acceptable alternative to an in-person office visit as determined by satisfaction with the program and the amount of further medical management required by the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over 18 and under 75 years of age undergoing elective primary orthopaedic surgery at Thomas Jefferson University Hospital, Rothman Orthopaedic Specialty Hospital or Methodist Hospital who have the capability to utilize a telecommunications platform (computer, tablet or similar device at home with a webcam, microphone and access to high-speed internet).

Exclusion Criteria:

1. Subjects who are unable to access the telemedicine platform or who are uncomfortable with following up in this fashion
2. Subjects who are unable or unwilling to provide post-operative radiographs electronically or who are unable or unwilling to obtain them
3. Subjects with workman's compensation or automotive claims or other ongoing litigation
4. Subjects that are unable or unwilling to consent for enrollment
5. Patients under the age of 18 years
6. Pregnant or breastfeeding women
7. Patients undergoing surgery for tumor, trauma or infection or who require revision or staged procedures
8. Patients without English-language proficiency
9. Patients with unforeseen intra-operative or perioperative complications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2017-10-06 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction: Likert Score | 2 mont post-operative period following surgery
  Likert Score self-reported patient satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States